CLINICAL TRIAL: NCT06260644
Title: Evaluation of Using Self-adhering Flowable Resin Composite Versus Conventional Nano-filled Flowable Resin Composite in Repairing Old Defective Resin Composite Restorations Over 18 Months Follow up. (A Randomized Clinical Trial)
Brief Title: Evaluation of Using Self-adhering Flowable Resin Composite in Repairing Old Defective Resin Composite Restorations Over 18 Months Follow up. (A Randomized Clinical Trial)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Soha Sayed Hosny, masters degree student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Repairing defective composite
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Occlusal Caries
Keywords: flowable resin composite

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: double ( participants, outcomes assessor) participants and both assessors will be blind to the type of material used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional flowable nano filled resin composite (Active Comparator): Repairing the old defective class I composite restoration by conventional nano filled flowable resin composite.
  Interventions: Procedure: VertiseTM flowable composite (Kerr,USA)
- Self adhesive flowable resin composite (Experimental): Repairing the old defective class I composite restoration by self adhering flowable resin composite.
  Interventions: Procedure: VertiseTM flowable composite (Kerr,USA)

INTERVENTIONS:
Procedure: VertiseTM flowable composite (Kerr,USA) — self adhesive flowable resin composite restoration.

SUMMARY:
This research proposal is evaluating the clinical performance of using self-adhering flowable resin composite in repairing old occlusal defective resin composite versus conventional flowable resin composite restoration over 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18-35 y)
* patients with defective resin composite class I restorations that need repair.
* dental motivated patients who attends regularly.
* Vital posterior teeth with repairable defective resin composite class I restorations.
* Localized marginal defect or marginal staining FDI 3& 4.
* Teeth with no or minimum mobility & healthy peridontium.
* No history of any irreversible pulpal pain or necrosis in the teeth to be restored.

Exclusion Criteria:

* • Patients with defective restorations that dictate replacement

  * Uncooperative behavior limits the isolation techniques throughout the procedure.
  * Presence of parafunctional habits.
  * Patient with history of systemic medical disease, or any other serious relevant problem.
  * High caries risk patients. Periodontal disease that may affect the prognosis of the restoration or the tooth itself.
  * Fractured or visibly cracked teeth.
  * Symptoms of any pulp pathosis.
  * Defective resin composite restorations that dictate replacement.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Restoration clinical performance using FDI criteria | assessment will be done after the treatment then 6 months, 12 months and18 months.
  FDI criteria mechanical parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No